CLINICAL TRIAL: NCT05651061
Title: To Evaluate the Safety, PK/PD and Immunogenicity of SS109 in Hemophilia Patients With Blood Coagulation Factor Ⅷ or Ⅸ Inhibitors After Single Administration, Open Label, Dose Escalation, and Multicenter Phase I Clinical Trial
Brief Title: A Phase I of SS109 in Hemophilia A or and B With Inhibitors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Gensciences lnc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTR20222792
Record Dates: First submitted 2022-11-29; First posted 2022-12-14 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-05

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia B With Inhibitor; Factor VII Deficiency
MeSH Terms: conditions — Factor VII Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose cohorts (Experimental): Dose cohorts were designed to evaluate the safety, immunogenicity and PK/PD.
  Interventions: Biological: SS109

INTERVENTIONS:
Biological: SS109 — 27 patients are enrolled in cohorts ,and will continue to be followed up until 28 days after SS109 administration for evaluating safety, PK/PD and immunogenicity.

SUMMARY:
This phase I study aims to evaluate the safety, PK/PD and immunogenicity of SS109 in hemophilia A or and B with inhibitors. Twenty -seven patients are enrolled in study, and divided into five dose cohorts, from 30μg/kg to 360μg/kg. Dose 1 cohort enrolls three patients, each other dose cohorts enroll six patients. All patients included in the study will continue to be followed up until 28 days after SS109 administration.

DETAILED DESCRIPTION:
This study is an open label, dose escalation, multicenter clinical trial. The study sets up a science review committee to assess the dose escalation. Serial blood samples for PK/PD analysis will be taken up to 72 hours after SS109 injection. Patients safety will be routinely monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age was 18 to 65 years old，when signing the informed consent form, male;
2. Clinical diagnosis of hemophilia A or B (previous or screening period FⅧ activity level≤ 1% or FⅨ activity level≤ 2%), and there is one of the following conditions:

   * FⅧ or FⅨ inhibitor level ≥ 5Bu/mL during screening period;
   * During the screening period, the level of FⅧ and FⅨ inhibitors was less than 5 Bu/mL and more than 0.6 Bu/mL, but had a high response to factor Ⅷ or IX injection (such as, the patient had a positive history of FⅧ/FⅨ inhibitors, and then the inhibitor level is ≥ 5Bu/mL, after the second infusion of FⅧ/FⅨ);
3. No active bleeding symptoms before the first injection;
4. Patients can comply with the requirements of the protocol and be willing to complete the study as planned and provide biological samples for test;
5. Be able to understand the procedures and methods of this clinical trial. The patient voluntarily participates and signs by himself or by the impartial witness

Exclusion Criteria:

1. Patients with known history of hypersensitivity to the investigational drug preparation and any of its components;
2. There was hypersensitivity or anaphylaxis after FⅦ or IgG2 injection treatment in the past;
3. Patients with FⅦ inhibitor positive or with FⅦ inhibitor positive history in screening period;
4. Severe anemia (hemoglobin < 60g/L);
5. Platelet count < 100 × 109/L；
6. Patients with abnormal liver and kidney functions: alanine aminotransferase (ALT) or aspartate aminotransferase (AST)≥ 2.5 times the upper limit of normal value (ULN), or total bilirubin ≥ 1.5 times ULN; or blood creatinine (Cr) ≥ 1.5 times;
7. One or more tests are positive, such as HBsAg, HCV antibody, anti-human immunity for HIV antibody and anti-treponema pallidum specific antibody (TPHA);
8. Except for hemophilia A or B, the coagulation indexes of any other bleeding disease or other diseases are obviously different(such as platelet disease, vitamin K deficiency, etc.);
9. History or symptoms of any previous arterial or venous thromboembolism event (such as atherosclerosis, myocardial infarction, ischemic stroke, transient ischemic attack, deep vein thrombosis or pulmonary hypertension, pulmonary embolism), or patients with history of disseminated intravascular coagulation (DIC);
10. Suffered from serious heart disease, such as unstable angina, congestive heart failure (New York Heart Association, ≥ Grade III), severe arrhythmia (QTc interval>450ms, corrected by Fridericia formula), hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 95 mmHg) not controlled by treatment;
11. Receive any product containing FⅦ or FⅦa (plasma derived or recombinate) within 48 hours before the first injection;
12. Receive any product containing FⅧ (plasma derived or recombinate) within 72 hours before the first injection; or receive any product containing FIX (plasma derived or recombinate) within 96 hours before administration;
13. Patients have used any anticoagulant, anti-fibrinol solvent, chemical, biological products or traditional Chinese medicine that affect platelet function within one week before the first injection or need to use any anticoagulant, anti-fibrinol solvent during PK/PD period, including non-steroidal anti-inflammatory drugs (NSAIDs) such as aspirin;
14. Patients have received immunomodulator (such as gamma globulin α- Interferon and prednisone>10mg/d [and>7 days] or similar drugs, except antiretroviral drugs);
15. Patients who received whole blood or plasma treatment within 2 weeks before the first injection;
16. Patients who have received vaccines within 4 weeks or planned to be vaccinated during the trial before the first injection;
17. Major surgery (such as orthopedic surgery and abdominal surgery) was performed within 1 month before the first injection, or planned to undergo surgery during the study;
18. Patients who have been selected into other clinical trials within 1 month before the first injection;
19. Patients with a history of drug abuse or alcohol abuse (alcohol abuse standard: male with a long-term alcohol consumption history of more than 5 years, equivalent to alcohol ≥ 40g/d, ≥ 20g/d for women, or a history of heavy drinking within 2 weeks, with the equivalent alcohol volume > 80g/d.
20. Patients suffering from mental illness or obvious mental disorder, or incapacity and lack of cognition caused by other reasons
21. A birth plan or sperm donation plan from the study to 3 months after the study, or patients are unwilling to take contraceptive measures (such as condoms, diaphragms, intrauterine devices, etc.);
22. A disease with clinical significance or other reasons that the researcher thinks patients are not suitable for participating in this clinical trial (if patients cannot benefit from clinical trials);
23. The investigator considers patients with poor compliance, and patients will be impossible to evaluate the efficacy or accomplish the course of treatment and follow-up.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse event/serious adverse event/specical interest adverse event(AE/SAE/AESI) | Up to 28 days after SS109 injected
  AE/SAE/AESI is any untoward clinical signs, symptoms or outcomes
Number of patients with positive FVII inhibitor, anti- drug antibody (ADA) | Up to 28 days after SS109 injected
  Number of patients with positive FVII inhibitor, anti drug antibody (ADA)

SECONDARY OUTCOMES:
t½ | Up to 72 hours after SS109 injected
  Half-life
Cmax | Up to 72 hours after SS109 injected
  Maximum concentration
Tmax | Up to 72 hours after SS109 injected
  Time to reach maximum concentration
AUC0-last | Up to 72 hours after SS109 injected
  Area under the curve from 0 to last
AUC0-72 | Up to 72 hours after SS109 injected
  Area under the curve from 0 to 72 hour
AUC0-∞ | Up to 72 hours after SS109 injected
  Area under the curve from 0 to ∞
CL | Up to 72 hours after SS109 injected
  Clearance
Vd | Up to 72 hours after SS109 injected
  Volume of distribution
MRT | Up to 72 hours after SS109 injected
  Mean residence time
IR | Up to 72 hours after SS109 injected
  Incremental recovery rate

OTHER OUTCOMES:
PT | Up to 72 hours after SS109 injected
  Prothrombin time
aPTT | Up to 72 hours after SS109 injected
  activated partial thromboplastin time
TGA | Up to 72 hours after SS109 injected
  thrombin generation test
TAT | Up to 72 hours after SS109 injected
  thrombin antithrombin complex

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, Principal Investigator — Hematology Hospital, Chinese Academy of Medical Sciences
Locations (10):
- China (10):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Henan Provincial Cancer Hospital, Zhengzhou, Henan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xi'an Central Hospital, Xi’an, Shanxi
  - Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No